CLINICAL TRIAL: NCT00933335
Title: Fludarabine Monophosphate Followed by Iodine I 131 Tositumomab for Untreated Low-grade and Follicular Non-Hodgkin's Lymphoma
Brief Title: Study of Safety and Efficacy of a Sequential Regimen Consisting of Three Cycles of Fludarabine Followed by Tositumomab and Iodine I 131 Tositumomab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 393229/023
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

ARMS (1):
- Single Arm (Experimental): Patients will first receive an abbreviated course of three cycles of fludarabine (25 mg/m2 for 5 days every 5 weeks). Iodine I 131 tositumomab will be initiated 6 to 8 weeks after completion of fludarabine. Patients will undergo dosimetry studies to determine the appropriate patient-specific activity of iodine I 131 tositumomab required to deliver a fixed dose of 75 cGy. The dose will be attenuated to 65 cGy for patients with platelet counts between 100,000 and 150,000/micoliter.
  Interventions: Biological: Tositumomab and Iodine I 131 Tositumomab

INTERVENTIONS:
Biological: Tositumomab and Iodine I 131 Tositumomab — Tositumomab and Iodine I 131 Tositumomab

SUMMARY:
This is a single-arm, single institution, phase II study of fludarabine monophosphate followed by Iodine I 131 Tositumomab for patients with previously untreated, advanced-stage (stage III or IV) low-grade, transformed low-grade and follicular non-Hodgkin's lymphoma. The primary objective of the study will be to evaluate the safety of this treatment combination and the secondary endpoint will be to evaluate efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be age 18 years or older.
* Patients must have a histologically-confirmed diagnosis of low-grade or follicular non-Hodgkin's B-cell lymphoma.
* Patients must have Ann Arbor stage III or IV extent of disease after completing staging.
* Patients must have bi-dimensionally measurable disease. At least one lesion must have both perpendicular diameters > 2 cm.
* Patients must have evidence that their tumor expresses the CD20 antigen by immunohistochemistry or flow cytometry.
* Patients must have no previous treatment for NHL.
* Patients must have a Karnofsky performance status of at least 60% and an anticipated survival of at least 3 months.
* Patients must have absolute granulocyte count greater than or equal to 1500 cells/mm3 and a platelet count > 100,000 cells/mm3 within 14 days of study entry and not require sustained support with hematopoietic cytokines or transfusion of blood products.
* Patients must have adequate renal and hepatic function.
* Patients must sign IRB approved informed consent form(s) prior to study entry.

Exclusion Criteria:

* Patients who received systemic steroids within 1 week of study entry, except patients on maintenance steroid therapy for a non-cancerous disease.
* Patients with evidence of active infection requiring intravenous antibiotics at the time of study entry.
* Patients with New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation.
* Patients with known HIV Infection.
* Patients with known brain or leptomeningeal metastases.
* Patients who are pregnant or nursing. Patients of childbearing potential must undergo a pregnancy test at screening and on the day fludarabine treatment is started. Treatment is not to be administered until a negative result is obtained. Males and females must agree to use effective contraception for 6 months following the iodine I 131 tositumomab therapy.
* Patients with prior malignancy other than lymphoma, except for adequately-treated skin cancer in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years.
* Patients with hypersensitivity to fludarabine.
* Patients who are receiving either approved or non-approved (through another protocol) anti-cancer drugs or biologics.
* Patients who are HAMA positive.
* Patients with previous allergic reaction to iodine. This does not include reacting to intravenous iodine containing contrast materials.

Inclusion Criteria for Iodine I 131 Tositumomab Therapy

* Patients who completed 3 cycles of fludarabine.
* Patients must have absolute granulocyte count ≥ to 1500/mm3, platelet count of ≥ 100,000/mm3 (≥ 150,000/mm3 if > 25% bone marrow involvement at restaging), and not require sustained support with hematopoietic cytokines or transfusions with blood products.
* Patients must have adequate renal and hepatic function.

Exclusion criteria for Antibody Therapy

* Patients with active obstructive hydronephrosis.
* Patients with evidence of active infection requiring intravenous antibiotics.
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1998-08; Primary Completion 2009-12 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Leonard JP, Coleman M, Kostakoglu L, Chadburn A, Cesarman E, Furman RR, Schuster MW, Niesvizky R, Muss D, Fiore J, Kroll S, Tidmarsh G, Vallabhajosula S, Goldsmith SJ. Abbreviated chemotherapy with fludarabine followed by tositumomab and iodine I 131 tositumomab for untreated follicular lymphoma. J Clin Oncol. 2005 Aug 20;23(24):5696-704. doi: 10.1200/JCO.2005.14.803. PMID 16110029
- See also: Leonard JP, Coleman M, Kostakoglu L, Chadburn A, Cesarman E, Furman R, et al. Abbreviated Chemotherapy with Fludarabine Followed by Tositumomab and Iodine I 131 Tositumomab for Untreated Follicular Lymphoma. J Clin Oncol 2005;23:5696-5704 — http://jco.ascopubs.org/cgi/content/full/23/24/5696
- Available data/document: Dataset Specification: 393229/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 393229/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 393229/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 393229/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 393229/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 393229/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 393229/023 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received fludarabine in the first study phase. Upon completion of this phase, if they met the appropriate criteria, they began the first of 2 phases of radioimmunotherapy: Phase 1, dosimetric dose (DD), administered 6 weeks after Day 1 of the third fludarabine cycle; Phase 2, therapeutic dose, administered 7-14 days after the DD.
Groups:
- Received Less Than 3 Cycles of Fludarabine: Participants received less than 3 cycles of intravenous (IV) fludarabine monophosphate (25 milligrams/meter^2/day [mg/m^2/day]) for 5 days every 5 to 6 weeks.
- Fludarabine (3 Cycles); TST and Iodine I 131 TST: Participants (par.) received 3 cycles of IV fludarabine (FL) monophosphate (25 mg/m^2/day) for 5 days every 5-6 weeks. After receiving FL, par. meeting criteria received the dosimetric dose (DD), administered 6-8 weeks after the 3rd cycle of FL. IV administration of unlabeled tositumomab (TST) (450 mg) was infused over 1 hour (hr) prior to a 30 minute infusion of 35 mg TST trace labeled with 5 millicurie (mCi) iodine I 131. Par. received >=3 doses (4 drops by mouth [DBM], 3 times a day [TID]) of a saturated solution of potassium iodide (KI), 3 doses (20 DBM, TID) of Lugol's solution, or KI tablets (130 mg BM, once a day) >=24 hrs prior to administration of the DD and continued daily for 14 days after the therapeutic dose (TD), administered 7-14 days after the DD. The TD was an IV infusion of 450 mg TST over 1 hr, followed by infusion of 35 mg of TST radiolabeled with iodine I 131 to deliver the appropriate total body dose of 75, 65, or 45 centigray (cGy) over 20 minutes.
Period: Overall Study
Arm/Group | Received Less Than 3 Cycles of Fludarabine | Fludarabine (3 Cycles); TST and Iodine I 131 TST
Started | 2 | 36 (35/36 participants who received 3 cycles of fludarabine later received a DD and TD of TST/I 131 TST.)
Completed | 0 | 20
Not Completed | 2 | 16
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Progressive Disease | 0 | 11
Not completed — Didn't Meet Criteria for TST/I 131 TST | 0 | 1
Not completed — Co-morbid Illness | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Received Less Than 3 Cycles of Fludarabine | Fludarabine (3 Cycles); TST and Iodine I 131 TST | Total
Number analyzed (Participants) | 2 | 36 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (11.3) | 51.2 (13.4) | 51.7 (13.4)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 16 | 17
  Male | 1 | 20 | 21
Race/Ethnicity, Customized [Number; unit: participants]
  White | 2 | 34 | 36
  Hispanic | 0 | 1 | 1
  Black | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and does not necessarily have to have a causal relationship (association) with this treatment. Therefore, an AE was any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not it was considered to be related to the medicinal product. Laboratory abnormalities were recorded as AEs only if they were associated with clinical sequelae and/or required an intervention.
Time Frame: First day of fludarabine cycle 1 to day prior to TST and iodine I 131 TST dosimetric dose (DD) (Week -16 to Week 1); Day of TST and iodine I 131 TST DD to database release (Week 1 to Week 520)
Population: Intent-to-Treat (ITT)-Exposed Population: all participants who were enrolled into the study and who received at least 1 dose of fludarabine. The data are presented for the subgroup of the ITT-Exposed Population for those participants who received the dosimetric and therapeutic dose of TST/I 131 TST.
Measure: Number; unit: participants
Groups:
- Fludarabine: Participants received 3 cycles of intravenous (IV) fludarabine monophosphate (25 mg/m^2/day) for 5 days every 5 to 6 weeks.
- TST and Iodine I 131 TST: The dosimetric dose (DD) was administered 6 to 8 weeks after the third cycle of fludarabine. IV administration of unlabeled tositumomab (TST) (450 mg) was infused over 1 hour (hr) prior to a 30 minute infusion of 35 mg TST trace labeled with 5 millicurie (mCi) iodine I 131. Participants received at least 3 doses (4 drops by mouth, 3 times a day [TID]) of a saturated solution of potassium iodide (KI), 3 doses (20 drops by mouth, TID) of Lugol's solution, or KI tablets (130 mg by mouth, once a day) 24 hrs or more prior to administration of the DD and continued daily for 14 days following the therapeutic dose (TD). The TD was administered 7 to 14 days after the dosimetric dose. The TD was an IV infusion of 450 mg TST over 1 hour, followed by infusion of 35 mg of TST radiolabeled with iodine I 131 to deliver the appropriate total body dose of 75, 65, or 45 centigray (cGy) over 20 minutes.
- Fludarabine/TST and Iodine I 131 TST (Combined Regimen): Participants received 3 cycles of IV fludarabine monophosphate (25 mg/m^2/day) for 5 days every 5 to 6 weeks. The DD was administered 6 to 8 weeks after the third cycle of fludarabine. IV administration of unlabeled TST (450 mg) was infused over 1 hr prior to a 30 minute infusion of 35 mg TST trace labeled with 5 mCi iodine I 131. Participants received at least 3 doses (4 drops by mouth, TID) of a saturated solution KI, 3 doses (20 drops by mouth, TID) of Lugol's solution, or KI tablets (130 mg by mouth, once a day) 24 hrs or more prior to administration of the DD and continued daily for 14 days following the TD. The TD was administered 7 to 14 days after the dosimetric dose. The TD was an IV infusion of 450 mg TST over 1 hour, followed by infusion of 35 mg of TST radio labeled with iodine I 131 to deliver the appropriate total body dose of 75, 65, or 45 cGy over 20 minutes.
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 38 | 35 | 38
participants | 33 | 34 | 38

2. Primary Outcome: Number of Participants With Any Treatment-related Adverse Event (TRAE)
Description: All noxious and unintended responses to a study treatment related to any dose were considered as TRAEs. A response to a study treatment indicates that a causal relationship between a study drug and an adverse event was at least a reasonable possibility, i.e., the relationship cannot be ruled out.
Time Frame: First day of fludarabine cycle 1 to day prior to TST and iodine I 131 TST DD (Week -16 to Week 1); Day of TST and iodine I 131 TST DD to database release (Week 1 to Week 520)
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 38 | 35 | 38
participants | 32 | 34 | 38

3. Primary Outcome: Number of Participants With Any Grade 3 or Grade 4 Adverse Event
Description: Adverse events were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No adverse event or within normal limits; 1 = Mild adverse event; 2 = Moderate adverse event; 3 = Severe and undesirable adverse event; 4 = Life-threatening or disabling adverse event; 5 = Death related to adverse event.
Time Frame: as for outcome 2
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 38 | 35 | 38
participants | 17 | 30 | 34

4. Primary Outcome: Number of Participants With Any Treatment-related Grade 3 or Grade 4 Adverse Event
Description: All of the treatment-related grade 3 (severe and undesirable) and grade 4 (life-threatening or disabling) adverse events experienced by the participants were recorded.
Time Frame: as for outcome 2
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 38 | 35 | 38
participants | 16 | 30 | 34

5. Primary Outcome: Number of Participants With Any Serious Adverse Event (SAE)
Description: An SAE was defined as any event occurring at any dose that results in any of the following outcomes: death, a life threatening adverse drug experience (at immediate risk of death from the experience as it occurred), inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered to be a serious adverse drug experience when based upon appropriate medical judgment.
Time Frame: as for outcome 2
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 38 | 35 | 38
participants | 2 | 7 | 8

6. Primary Outcome: Number of Participants With Any Treatment-related SAE
Description: All of the treatment-related SAEs experienced by the participants were recorded.
Time Frame: as for outcome 2
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 38 | 35 | 38
participants | 0 | 7 | 7

7. Primary Outcome: Number of Participants With the Indicated Grade 3 and Grade 4 AEs
Description: AEs were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No AE or within normal limits; 1 = Mild AE; 2 = Moderate AE; 3 = Severe and undesirable AE; 4 = Life-threatening or disabling AE; 5 = Death related to AE. mm, millimeters; mm^3, millimeters cubed. Grade 3 and Grade 4 AEs are reported to focus on the most severe AEs.
Time Frame: as for outcome 2
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 38 | 35 | 38
participants
  Absolute neutrophil count <1000 cells/mm^3 | 11 | 27 | 31
  White blood cell count <2000 cells/mm^3 | 12 | 26 | 30
  Platelet count <50000 cells/mm^3 | 3 | 17 | 19
  Hemoglobin <8.0 grams/deciliter | 1 | 10 | 11
  Neutropenia | 7 | 2 | 9
  Anaemia | 1 | 3 | 4
  Leukopenia | 1 | 3 | 4
  Thrombocytopenia | 1 | 2 | 3
  Febrile neutropenia | 0 | 2 | 2
  Myelodysplastic syndrome | 0 | 2 | 2
  Acute myeloid leukaemia | 0 | 1 | 1
  Chronic myelomonocytic leukaemia | 0 | 1 | 1
  Prostate cancer | 0 | 1 | 1
  Squamous cell carcinoma | 0 | 1 | 1
  Nausea | 1 | 1 | 2
  Arrhythmia | 1 | 0 | 1
  Cardiac failure congestive | 1 | 0 | 1
  Left ventricular dysfunction | 1 | 0 | 1
  Myocardial infarction | 1 | 0 | 1
  Autoimmune thyroiditis | 0 | 1 | 1
  Pyrexia | 1 | 0 | 1
  Headache | 0 | 1 | 1
  Dyspnoea | 1 | 0 | 1

8. Primary Outcome: Number of Participants With the Indicated Treatment-related AEs Experienced by at Least 10% of Participants in the Combined Regimen
Description: as for outcome 2
Time Frame: as for outcome 2
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 38 | 35 | 38
participants
  Absolute neutrophil count <1000 cells/mm^3 | 11 | 27 | 31
  White blood cell count <2000 cells/mm^3 | 12 | 26 | 30
  Platelet count <50000 cells/mm^3 | 3 | 17 | 19
  Hemoglobin <8.0 grams/deciliter | 1 | 10 | 11
  Fatigue | 7 | 11 | 16
  Pyrexia | 8 | 10 | 14
  Asthenia | 5 | 5 | 9
  Chills | 3 | 3 | 6
  Nausea | 12 | 9 | 18
  Vomiting | 2 | 5 | 7
  Rash | 6 | 2 | 8
  Ecchymosis | 1 | 4 | 5
  Headache | 3 | 6 | 8
  Dizziness | 0 | 5 | 5
  Neutropenia | 11 | 2 | 12
  Anaemia | 2 | 9 | 10
  Leukopenia | 3 | 3 | 5
  Myalgia | 1 | 4 | 5
  Arthralgia | 0 | 4 | 4
  Cough | 5 | 10 | 14
  Nasal congestion | 4 | 6 | 8
  Dyspnoea | 2 | 5 | 6
  Oropharyngeal pain | 2 | 4 | 6
  Rhinorrhoea | 2 | 2 | 4
  Sinusitis | 2 | 3 | 5
  Nasopharyngitis | 1 | 3 | 4
  Decreased appetite | 6 | 4 | 10
  Insomnia | 2 | 2 | 4
  Palpitations | 1 | 3 | 4

9. Primary Outcome: Number of Participants Who Were Negative for Human Anti-murine Antibodies (HAMA) at Baseline (Study Entry) But Positive or Negative at Weeks 12 and 25 and at Months 12, 18, and 24
Description: The administration of murine antibodies may form HAMA. A HAMA assay was performed using the ImmunoSTRIP HAMA IgG enzyme-linked immune absorbent assay by a central laboratory (Covance Classic Laboratory Services, Indianapolis, IN). Fludarabine, a known immunosuppressant, might decrease HAMA production in addition to reducing bone marrow involvement. To be "positive," a participant had to have a positive HAMA assessment at any follow-up visit (Weeks 12 and 25; Months 12, 18, and 24).
Time Frame: Day 1 to Day 730 (24 Months) after receiving the dosimetric dose
Population: ITT-Exposed Population: participants who were evaluable for HAMA (those who did not have a positive HAHA level at Baseline) and those who received dosimetric and therapeutic doses were evaluated.
Measure: Number; unit: participants
Groups:
- Fludarabine/TST and Iodine I 131 TST: Participants received 3 cycles of IV fludarabine monophosphate (25 mg/m^2/day) for 5 days every 5 to 6 weeks. The DD was administered 6 to 8 weeks after the third cycle of fludarabine. IV administration of unlabeled TST (450 mg) was infused over 1 hr prior to a 30 minute infusion of 35 mg TST trace labeled with 5 mCi iodine I 131. Participants received at least 3 doses (4 drops by mouth, TID) of a saturated solution KI, 3 doses (20 drops by mouth, TID) of Lugol's solution, or KI tablets (130 mg by mouth, once a day) 24 hrs or more prior to administration of the DD and continued daily for 14 days following the TD. The TD was administered 7 to 14 days after the dosimetric dose. The TD was an IV infusion of 450 mg TST over 1 hour, followed by infusion of 35 mg of TST radio labeled with iodine I 131 to deliver the appropriate total body dose of 75, 65, or 45 cGy over 20 minutes.
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 32
participants
  Positive | 2
  Negative | 30

10. Primary Outcome: Time to HAMA Positivity From the First TST/I 131 TST Dosimetric Dose for the Participants Achieving HAMA Positivity
Description: Kaplan-Meier estimates of the time to HAMA positivity (days from the first fludarabine dose) was determined for participants who converted to HAMA positivity.
Time Frame: Day 1 to Day 730 (24 Months) after receiving the dosimetric dose
Population: ITT-Exposed Population: participants who received dosimetric and therapeutic doses and those who were converted to HAMA positivity were evaluated.
Measure: Number; unit: days
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 2
days
  Participant 1 | 184 (7.8)
  Participant 2 | 195

11. Primary Outcome: Number of Participants With Elevated Thyroid-Stimulating Hormone (TSH) Levels at Baseline (Study Entry) and Weeks 25, 52, 78, 104, 130, 156, 182, 208, 234, 260, 286, 312, 364, 416, 468, and 512
Description: The number of participants with elevated TSH levels is reported. An elevated TSH level indicates that an insufficient amount of the thyroid hormone is being produced. Insufficient thyroid hormone production is known as hypothyroidism. The normal range of TSH is between 0.2 and 6.1 milliunits per liter (mU/L).
Time Frame: Baseline (Week -16) and Weeks 25, 52, 78, 104, 130, 156, 182, 208, 234, 260, 286, 312, 364, 416, 468, and 512
Population: ITT-Exposed Population: baseline TSH levels were determined for 36 participants. Of 35 participants who received the dosimetric and therapeutic doses of TST/I-131 TST, 2 had elevated TSH at baseline, and 33 were assessed for developing elevated TSH.
Measure: Number; unit: participants
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 35
participants
  Baseline (Week -16), n=35 | 2
  Week 25, n=33 | 3
  Week 52, n=33 | 1
  Week 78, n=33 | 4
  Week 104, n=33 | 3
  Week 130, n=33 | 1
  Week 156, n=33 | 0
  Week 182, n=33 | 0
  Week 208, n=33 | 0
  Week 234, n=33 | 0
  Week 260, n=33 | 0
  Week 286, n=33 | 0
  Week 312, n=33 | 1
  Week 364, n=33 | 1
  Week 416, n=33 | 0
  Week 468, n=33 | 0
  Week 512, n=33 | 0

12. Primary Outcome: Number of Participants With Thyroid Medication Use Prior to the Therapeutic Dose
Description: Thyroid medication included any prescribed medication for the treatment of thyroid dysfunction.
Time Frame: Baseline (study entry; Week -16) and Week 2 to Week 3 (prior to the therapeutic dose)
Population: ITT-Exposed Population: all participants who received dosimetric and therapeutic doses were evaluated.
Measure: Number; unit: participants
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 35
participants | 0

13. Primary Outcome: Time to Nadir for Hematological Parameters: Absolute Neutrophil Count (ANC), Hemoglobin, and Platelets
Description: Nadir was defined as the lowest laboratory value recorded up to 120 days following the therapeutic dose (or dosimetric dose for participants who did not receive the therapeutic dose).
Time Frame: up to 120 days following the therapeutic dose (or dosimetric dose for participants who did not receive the therapeutic dose)
Population: ITT-Exposed Population: all participants who received the dosimetric dose were evaluated.
Measure: Median (Full Range); unit: days
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 35
days
  ANC | 48 [36 to 90]
  Hemoglobin | 50 [28 to 87]
  Platelets | 36 [22 to 48]

14. Primary Outcome: Nadir Values for Absolute Neutrophil Count (ANC)
Description: as for outcome 13
Time Frame: as for outcome 13
Population: ITT-Exposed Population: only the 35 participants who received the dosimetric dose were evaluated.
Measure: Median (Full Range); unit: 10^3/mm^3
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 35
10^3/mm^3 | 0.8 [0 to 4]

15. Primary Outcome: Nadir Values for Hemoglobin
Description: as for outcome 13
Time Frame: as for outcome 13
Population: ITT-Exposed Population: only the 35 participants who received the dosimetric dose were evaluated.
Measure: Median (Full Range); unit: g/dL
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 35
g/dL | 10.7 [6 to 15]

16. Primary Outcome: Nadir Values for Platelet Count
Description: as for outcome 13
Time Frame: as for outcome 13
Population: ITT-Exposed Population: only the 35 participants who received the dosimetric dose were evaluated.
Measure: Median (Full Range); unit: 10^3/microliter
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 35
10^3/microliter | 53 [4 to 126]

17. Primary Outcome: Number of Participants With Any Grade 3 or Grade 4 Toxicity (AE) for Hematological Parameters (Absolute Neutrophil Count [ANC], Hemoglobin, and Platelets)
Description: Adverse events were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades (G): 0=No AE or within normal limits; 1=Mild AE; 2=Moderate AE; 3=Severe and undesirable AE; 4=Life-threatening or disabling AE; 5=Death related to AE. ANC (10^3/mm^3): G1=1.5 to <2.0, G2=1.0 to <1.5, G3=0.5 to < 1.0, G4=<0.5. Hemoglobin (g/dL): G1=10.0 to <12.0, G2=8.0 to <10.0, G3=6.5 to <8.0, G4=< 6.5. Platelets (10^3/microliter): G1=75 to <150, G2=50 to <75, G3=25 to <50, G4=<25.
Time Frame: as for outcome 1
Population: ITT-Exposed Population: all participants who received dosimetric and therapeutic doses were evaluated.
Measure: Number; unit: participants
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 35
participants
  ANC | 28
  Hemoglobin | 10
  Platelets | 17

18. Primary Outcome: Duration of Any Grade 3 or Grade 4 Toxicity for Hematological Parameters: Absolute Neutrophil Count (ANC), Hemoglobin, and Platelets
Description: as for outcome 17
Time Frame: as for outcome 1
Population: ITT-Exposed Population: all participants who received dosimetric and therapeutic doses were evaluated.
Measure: Median (Full Range); unit: days
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 35
days
  ANC | 31 [2 to 877]
  Hemoglobin | 16 [3 to 199]
  Platelets | 29 [2 to 83]

19. Primary Outcome: Number of Participants With Any Infection at Week 16 Post-Fludarabine Treatment and Week 13 Post-TST Treatment Detected by Laboratory Culture of Participant Sample or Investigator Report
Description: An infection is the colonization of a host organism by a parasite species. Infecting parasites seek to use the host's resources to reproduce, often resulting in disease. Colloquially, infections are usually considered to be caused by microscopic organisms or microparasites like viruses, bacteria, and viroids, although larger organisms such as macroparasites and fungi can also infect.
Time Frame: Week 16 Post-Fludarabine Treatment (Week -16 to Week 0); Week 13 Post-TST Treatment (Week 1 to Week 13)
Population: ITT-Exposed Population: all participants who received dosimetric and therapeutic doses were evaluated.
Measure: Number; unit: participants
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 35
participants
  Week 16 Post-Fludarabine Treatment | 11
  Week 13 Post-TST Treatment | 9

20. Primary Outcome: Number of the Indicated Type of Infection Reported by Investigator Based on Laboratory Testing at Week 16 Post-Fludarabine (Fl) Treatment and Week 13 Post-TST Treatment
Description: as for outcome 19
Time Frame: Week 16 Post-Fludarabine Treatment (Week -16 to Week 0); Week 13 Post-TST Treatment (Week 1 to Week 13)
Population: ITT-Exposed Population: all participants who received dosimetric and therapeutic doses and those who had an infection were evaluated. A single participant could have had more than one infection. The number analyzed in the category titles reflects the number of participants who had any infection.
Measure: Number; unit: number of infections
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 11
number of infections
  Week 16 Post-Fl treatment, Pneumonia, n=11 | 1
  Week 16 Post-Fl treatment, Other Infections, n=11 | 12
  Week 13 Post-TST Treatment, Pneumonia, n=9 | 0
  Week 13 Post-TST Treatment, Other Infections, n=9 | 9

21. Primary Outcome: Number of Participants With a Culture Obtained for Infection at Week 16 Post-Fludarabine (Fl) Treatment and Week 13 Post-TST Treatment
Description: Specimen samples of the body fluid are cultured for testing whether the infectious organism is present and grown in the culture media to assess the growth pattern of the organisms present in the specimen.
Time Frame: Week 16 Post-Fludarabine Treatment (Week -16 to Week 0); Week 13 Post-TST Treatment (Week 1 to Week 13)
Population: ITT-Exposed Population: all participants who received dosimetric and therapeutic doses and those who had an infection were evaluated.
Measure: Number; unit: participants
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 11
participants
  Week 16 Post-Fl treatment, n=11 | 2
  Week 13 Post-TST Treatment, n=9 | 1

22. Primary Outcome: Number of Participants With Positive Culture Results for Infections at Week 16 Post-Fludarabine (Fl) Treatment and Week 13 Post-TST Treatment
Description: The culture results could be positive or negative. The positive culture results indicates that the tested participant have the infection under investigation so therapeutic treatment with anti-infective is required.
Time Frame: Week 16 Post-Fludarabine Treatment (Week -16 to Week 0); Week 13 Post-TST Treatment (Week 1 to Week 13)
Population: ITT-Exposed Population: all participants who received dosimetric and therapeutic doses, those who had an infection, and from whom the cultures were obtained were evaluated.
Measure: Number; unit: participants
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 2
participants
  Week 16 Post-Fl treatment, n=2 | 0
  Week 13 Post-TST Treatment, n=1 | 0

23. Primary Outcome: Number of Participants With an Anti-infective Administered at Week 16 Post-Fludarabine (Fl) Treatment and Week 13 Post-TST Treatment
Description: Anti-infectives are capable of acting against infection, by inhibiting the spread of an infectious agent or by killing the infectious agent outright. Anti-infective is a general term that encompasses antibacterials, antibiotics, antifungals, antiprotozoans, and antivirals.
Time Frame: Week 16 Post-Fludarabine Treatment (Week -16 to Week 0); Week 13 Post-TST Treatment (Week 1 to Week 13)
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 11
participants
  Week 16 Post-Fl treatment, n=11 | 11
  Week 13 Post-TST Treatment, n=9 | 9

24. Primary Outcome: Number of Participants Who Received Any Supportive Care After Fludarabine Treatment and After TST Treatment
Description: Supportive care involves interventions that help the participants to achieve comfort but do not affect the course of a disease.
Time Frame: as for outcome 2
Population: ITT-Exposed Population: two participants who received less than 3 cycles of fludarabine did not receive TST treatment, and hence were not evaluated.
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST
Number analyzed (Participants) | 36 | 35
participants | 15 | 14

25. Primary Outcome: Number of Participants Receiving the Indicated Type of Supportive Care After Fludarabine Treatment and After TST Treatment
Description: Supportive care involves interventions that help the participants to achieve comfort but do not affect the course of a disease. Supportive care involved administration of granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GM-CSF), red blood cell (RBC) transfusions, erythropoietin, and platelet transfusions.
Time Frame: First day of fludarabine cycle 1 to day prior to TST/I 131 TST dosimetric dose (Week -16 to Week 1); Day of TST/I 131 TST dosimetric dose to database release (Week 1 to Week 520)
Population: ITT-Exposed Population: two participants who received less than 3 cycles of fludarabine did not receive TST treatment and were not evaluated.
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST
Number analyzed (Participants) | 36 | 35
participants
  G-CSF/GM-CSF | 10 | 10
  RBC transfusion | 8 | 7
  Erythropoietin | 7 | 7
  Platelet transfusion | 3 | 2

26. Secondary Outcome: Number of Participants With the Investigator-assessed Confirmed Responses of Complete Response (CR), Clinical Complete Response (CCR), and Partial Response (PR)
Description: CR: Complete resolution of disease-related (DR) radiological abnormalities; disappearance of non-Hodgkin's lymphoma-related signs/symptoms. CCR: Complete resolution of DR symptoms except for residual scar tissue. PR: 50% reduction in the sum of the products of the longest perpendicular diameters of measurable lesions with no new lesions. A confirmed response (resp.) (CR/CCR/PR) had to be confirmed by a consecutive resp. (>=28 days later) that was the same/better. Individual confirmed resp. data only counts that resp. confirmed by the same resp.; not all possible combinations are represented.
Time Frame: as for outcome 25
Population: ITT-Exposed Population. 2 participants (par.) who received <3 cycles of fludarabine (fl.) did not receive TST treatment and were not evaluated. Par. evaluable for response were those with >=1 assessment. Three par. were not evaluable for response. None of the responses could be confirmed after fl. treatment; thus, no data are reported for this arm.
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 38 | 32 | 35
participants
  Participants with CR, CCR, or PR | 0 | 30 | 32
  Participants with CR or CCR | 0 | 29 | 29
  Participants with PR | 0 | 1 | 2

27. Secondary Outcome: Number of Participants With the Investigator-assessed Unconfirmed Responses of Complete Response (CR), Clinical Complete Response (CCR), and Partial Response (PR)
Description: CR: Complete resolution of disease-related (DR) radiological abnormalities; disappearance of non-Hodgkin's lymphoma-related signs/symptoms. CCR: Complete resolution of DR symptoms except for residual scar tissue. PR: 50% reduction in the sum of the products of the longest perpendicular diameters of measurable lesions with no new lesions.
Time Frame: as for outcome 25
Population: ITT-Exposed Population. Participants (par.) evaluable for response were those with >= 1 response assessment. 2 of 38 par. who received <3 cycles of fludarabine withdrew from the study and were not evaluable for response. 35 of 38 par. received TST and I 131 TST treatment and were evaluated for response.
Measure: Number; unit: participants
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 36 | 35 | 36
participants
  Participants with CR, CCR, or PR | 32 | 32 | 36
  Participants with CR or CCR | 3 | 30 | 30
  Participants with PR | 29 | 2 | 6

28. Secondary Outcome: Number of Participants With Progression of Disease
Description: Progression of disease is defined as a 50% increase from nadir of the sum of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >2 cm in diameter per radiographic evaluation or >1 cm in diameter by physical examination. All participants without progression of disease were censored.
Time Frame: as for outcome 25
Population: ITT-Exposed Population: participants with confirmed response rates (CR, CCR, or PR) were evaluated.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 30 | 32
participants
  Progressed | 11 | 13
  Censored | 19 | 19

29. Secondary Outcome: Duration of Response for All Confirmed Responders
Description: Duration of response was defined as the time from the first documented response to the first documented disease progression. Partial Response (PR): 50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions with no new lesions. Responders are the participants with CR, or CCR, or PR.
Time Frame: as for outcome 25
Population: ITT-Exposed Population: all participants who received dosimetric and therapeutic doses and were classified as responders were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 30 | 32
months
  Participants with CR, CCR, or PR, n=30, 32 | NA [NA to NA] — The quartiles for duration of response are based on the Kaplan-Meier (KM) method. A median (50% quartile) was not reached because there were not enough events to reach a median on the KM curve. | NA [NA to NA] — The quartiles for duration of response are based on the Kaplan-Meier (KM) method. A median (50% quartile) was not reached because there were not enough events to reach a median on the KM curve.
  Participants with CR or CCR, n=29, 29 | NA [NA to NA] — The quartiles for duration of response are based on the Kaplan-Meier (KM) method. A median (50% quartile) was not reached because there were not enough events to reach a median on the KM curve. | NA [NA to NA] — The quartiles for duration of response are based on the Kaplan-Meier (KM) method. A median (50% quartile) was not reached because there were not enough events to reach a median on the KM curve.
  Participants with PR, n=1, 2 | 8.1 [NA to NA] — The procedure in SAS was not able to calculate the upper or lower limits of the confidence interval. | 9.4 [6.5 to 12.3]

30. Secondary Outcome: Number of Participants With Progressive Disease (PD)
Description: PD is defined as a 50% increase from nadir of the sum of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >2 cm in diameter per radiographic evaluation or >1 cm in diameter by physical examination.
Time Frame: as for outcome 25
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 35 | 38
participants | 19 | 21

31. Secondary Outcome: Time to Disease Progression or Death
Description: Time to progression is the time from the treatment start date to the first documented disease progression or death. Disease progression: 50% increase from nadir of the sum of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be >2 cm in diameter per radiographic evaluation or >1 cm in diameter by physical examination.
Time Frame: as for outcome 25
Population: ITT-Exposed Population. Participants with disease progression were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 19 | 21
months | 97.5 [26.9 to NA] — The procedure in SAS was not able to calculate the upper limit of the confidence interval. | 95.6 [30.9 to NA] — The procedure in SAS was not able to calculate the upper limit of the confidence interval.

32. Secondary Outcome: Number of Participants With a Treatment Failure
Description: Treatment failure is defined as the occurrence of treatment withdrawal, a decision to seek additional therapy, study removal, progression, alternative therapy for lymphoma, or death.
Time Frame: as for outcome 25
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 35 | 38
participants | 20 | 23

33. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from the treatment start date to the first occurrence of treatment withdrawal, a decision to seek additional therapy, study removal, progression, alternative therapy for lymphoma, or death.
Time Frame: as for outcome 25
Population: ITT-Exposed Population. Participants with treatment failure were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 20 | 23
months | 91.4 [26.3 to NA] — The procedure in SAS was not able to calculate the upper limit of the confidence interval. | 50.0 [29.6 to NA] — The procedure in SAS was not able to calculate the upper limit of the confidence interval.

34. Secondary Outcome: Number of Participants Who Died During Their Participation in the Study
Description: Participants who died during the study period were evaluated for the overall survival endpoint.
Time Frame: Day of TST/I 131 TST dosimetric dose to date of database release (Week 1 to Week 520); First day of fludarabine cycle 1 to date of database release (Week -16 to Week 520)
Population: ITT-Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Number analyzed (Participants) | 35 | 38
participants | 9 | 11

35. Secondary Outcome: Time to Death of Participants During Their Participation in the Study
Description: Time to death is defined as the time from the treatment start date to the date of death.
Time Frame: as for outcome 34
Population: ITT-Exposed Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST
Number analyzed (Participants) | 9 | 11
months | NA [NA to NA] — The quartiles for time to death are based on the Kaplan-Meier (KM) method. A median (50% quartile) was not reached because there were not enough events to reach a median on the KM curve. | NA [NA to NA] — The quartiles for time to death are based on the Kaplan-Meier (KM) method. A median (50% quartile) was not reached because there were not enough events to reach a median on the KM curve.

ADVERSE EVENTS:
Time Frame: All serious and non-serious adverse events (AEs) were reported up to Week 12 after the therapeutic dose. Thereafter, only AEs considered by the investigator to be possibly or probably associated with study treatment were required to be reported.
Groups:
- Fludarabine: Participants who received any number of cycles of IV fludarabine monophosphate (25 mg/m^2/day). Each cycle was administered for 5 days every 5 to 6 weeks.
Arm/Group | Fludarabine | TST and Iodine I 131 TST | Fludarabine/TST and Iodine I 131 TST (Combined Regimen)
Serious Adverse Events (participants affected / at risk) | 2/38 | 7/35 | 8/38
Other Adverse Events (participants affected / at risk) | 33/38 | 34/35 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine (N=38) | TST and Iodine I 131 TST (N=35) | Fludarabine/TST and Iodine I 131 TST (Combined Regimen) (N=38)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine (N=38) | TST and Iodine I 131 TST (N=35) | Fludarabine/TST and Iodine I 131 TST (Combined Regimen) (N=38)
Absolute neutrophil count (ANC) <1000 cells/mm^3 (Blood and lymphatic system disorders) | 11 | 27 | 31
White blood cells (WBC) <2000 cells/cmm (Blood and lymphatic system disorders) | 12 | 26 | 30
Platelets < 50000 cells/mm^3 (Blood and lymphatic system disorders) | 3 | 17 | 19
Hemoglobin <8.0 grams/deciliter (Blood and lymphatic system disorders) | 1 | 10 | 11
Fatigue (General disorders) | 7 | 11 | 16
Pyrexia (General disorders) | 9 | 10 | 15
Asthenia (General disorders) | 5 | 5 | 9
Chills (General disorders) | 3 | 3 | 6
Malaise (General disorders) | 1 | 1 | 2
Pain (General disorders) | 1 | 1 | 2
Axillary pain (General disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 1
Feeling abnormal (General disorders) | 1 | 0 | 1
Feeling cold (General disorders) | 1 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 1 | 1
Oedema (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 10 | 18
Vomiting (Gastrointestinal disorders) | 3 | 5 | 7
Constipation (Gastrointestinal disorders) | 2 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 1
Retching (Gastrointestinal disorders) | 0 | 1 | 1
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 2 | 8
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 4 | 5
Drug eruption (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 4 | 6 | 9
Somnolence (Nervous system disorders) | 1 | 7 | 8
Dizziness (Nervous system disorders) | 0 | 6 | 6
Sinus headache (Nervous system disorders) | 0 | 2 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 1
Sensory disturbance (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 11 | 2 | 12
Anaemia (Blood and lymphatic system disorders) | 2 | 9 | 10
Leukopenia (Blood and lymphatic system disorders) | 3 | 3 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 2 | 3 | 5
Nasopharyngitis (Infections and infestations) | 1 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3
Herpes zoster (Infections and infestations) | 0 | 2 | 2
Oral herpes (Infections and infestations) | 1 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 1
Device related infection (Infections and infestations) | 1 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 4 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2 | 4
Anxiety (Psychiatric disorders) | 1 | 3 | 3
Hallucination (Psychiatric disorders) | 1 | 0 | 1
Nightmare (Psychiatric disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 3 | 4
Tachycardia (Cardiac disorders) | 1 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma (Nervous system disorders) | 0 | 1 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1
Benign prostatic hyperplasi (Reproductive system and breast disorders) | 1 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 2 | 1 | 3
Hot flush (Vascular disorders) | 1 | 1 | 2
Pallor (Vascular disorders) | 0 | 1 | 1
Varicose vein (Vascular disorders) | 1 | 0 | 11
Hypothyroidism (Endocrine disorders) | 0 | 3 | 3
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 2 | 0 | 2
Azotaemia (Renal and urinary disorders) | 1 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 3 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 3
Blood pressure systolic decreased (Investigations) | 0 | 1 | 1
Heart rate increased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 1 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 1
Sinus operation (Surgical and medical procedures) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.